CLINICAL TRIAL: NCT02979795
Title: Translational Research in Identifying Molecular Mechanisms for Rectal Cancer Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Kun-San Clifford Chao, Cancer center, China Medical University Hospital
Other Study IDs: CMUH105-REC2-072
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Rectal Cancer; Chemoradiation
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Preoperative chemoradiotherapy — Preoperative chemoradiotherapy. 2.5 Gray/fraction (Total in 45-54 Gray)

SUMMARY:
Rectal cancer, comprised of 30% of overall colorectal cancer cohort, is one of the leading cancers of Taiwan. In patients with advanced disease, the standard of care is concurrent chemoradiotherapy (CCRT) before surgery. After CCRT, the abscopal effect, a phenomenon that localized radiation not only destroys local tumor but also inhibits the growth of tumor at the remote site, has been observed. This effect is believed to be associated with tumor immune response. In addition, other immune checkpoint molecules, such as Programmed cell death-1(PD-1), Programmed cell death ligand-1 (PD-L1), and Cytotoxic T-Lymphocyte Associated Protein 4 (CTLA-4), have been reported associated with therapeutic outcome. However, after CCRT, more than 50% of patients were still either having persistent disease or developed distant metastasis. To improve therapeutic outcome of patients with rectal cancer, this project, thus, aims at exploring the evolution of factors that may affect the abscopal effect and immune checkpoint functions in tissues and in blood before and after CCRT.

DETAILED DESCRIPTION:
For most patients, preoperative chemoradiotherapy results in clinically tumor regression, but the degree of response varies among patients. There are approximately 40-60% of LARC patients treated with CCRT achieve some degree of pathologic response. However, there is yet an effective method before the commencement of CCRT that can predict how patients will respond to CCRT and can subsequently render better survival. Identify patents who will benefit most from CCRT is crucial not only in lowering treatment-related morbidity and sustaining local control but also to improve survival rate in LARC.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer patients in China Medical University Hospital (Age limit: 20 yrs and older)

Exclusion Criteria:

* Pregnancy, Disabilities

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients in China Medical University Hospital (Age: 20 yrs and older)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Tumor regression rate | within 8 weeks after completion of chemoradiotherapy
  complete tumor regression rate(TRG) with tumor regression graded at at surgical resection at 8 weeks after completion of chemoradiotherapy

SECONDARY OUTCOMES:
Disease free survival | 5 year
Overall survival | 5 year
Local recurrence | 5 year
Distant metastasis | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Kan Sun Clifford Chao, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided